## Clinical Trial Statistical Analysis Plan

**Title:** Effects of Open-label Placebos Administered Through Telehealth on COVID-related

Stress, Anxiety, and Depression

Brief Title: Effects of Open-label Placebos on COVID-related Psychological Health

Study Sponsor: Michigan State University

## **Principle Investigator:**

Name: Jason S. Moser

Official Title: Professor of Psychology Affiliation: Michigan State University

Phone: 517-355- 2159 Email: jmoser@msu.edu

NCT Number: NCT05035550

Version Date: 1.22.21

## Statistical Analysis Plan

All analyses were conducted on SPSS version 26 (IBM, Armonk, NY). Prior to our primary analyses, we first interpolated missing data using a maximum likelihood estimation (MLE). Second, we conducted an independent sample t-test on baseline measures of each primary outcome measure to ensure that the control and open-label placebo group did not differ prior to the administration of the intervention.

The primary outcomes at the endpoint (reduction in COVID stress, perceived stress, anxiety, and depression) were calculated using change from baseline scores (endpoint minus baseline) with positive numbers indicating greater reduction in symptoms at endpoint. First, each primary outcome was submitted to a one-way analysis of covariance (ANCOVA), with group as the independent variable and the mean baseline score for each outcome measure submitted as a covariate to control for variability in baseline scores (Lembo et al., 2021; Van Breukelen, 2006). We reported outlier detection procedures and additional robust analyses in the Supplementary Materials. Effect sizes for pairwise comparisons were calculated using Cohen's d. Secondary outcomes were analyzed using descriptive statistics and t-tests. All significance tests were analyzed at p = .05.